CLINICAL TRIAL: NCT03096756
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study Designed to Compare the Safety and Pharmacokinetics of Orally Administered Superoxide Dismutase Mimetic GC4702 With Intravenously Administered Superoxide Dismutase Mimetic GC4419 (Part 1), With Assessment of Food Effect (Part 2), in Healthy Volunteers
Brief Title: A Study of the Safety, Tolerability and Pharmacokinetics of Orally-administered GC4702 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Collaborators: INC Research Australia Pty Ltd (Unknown); Nucleous Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GTO-001
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteer
Keywords: Oral Formulation; Food Effect; Superoxide Dismutase; Single Ascending Dose; GC4702; Bioavailability; Pharmacokinetics; Active Comparator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose Escalation GC4702 (Other): Serially increase dose escalation of orally formulated GC4702 or placebo (6:2 ratio), preceded by single dose of active comparator, GC4419 IV.
  Interventions: Drug: GC4702 dry powder; Drug: GC4702 lipid suspension; Other: GC4419 IV; Other: Placebo Dry Powder; Other: Placebo lipid suspension
- Part 2: Food Effect Study (Experimental): Following Part 1 dose find, single dose level of GC4702 administered under fasting for and fed condition.
  Interventions: Other: Fed Condition; Other: Fasting Condition; Drug: GC4702 lipid suspension - Part 2

INTERVENTIONS:
Drug: GC4702 dry powder — 5 mg GC4702 mixed with approximately 270 mg of Prosolv 90 LM - SMCC (siliconized microcrystalline cellulose). Planned dose levels of GC4702 encapsulated dry powder formulation are 50, 100, and 150 mg
  Arms: Part 1: Single Ascending Dose Escalation GC4702
Drug: GC4702 lipid suspension — 112 mg GC4702 mixed with Miglyol 812 plus 0.5% by weight BHA plus 1% by weight of Aerosil 200. Planned dose levels of GC4702 encapsulated lipid suspension formulation are 112, 224, and 336, 448, and 560 mg
  Arms: Part 1: Single Ascending Dose Escalation GC4702
Other: GC4419 IV — infused IV as a single dose of 27 mg (3 mL GC4419 at 9 mg/mL) in 247 mL normal (0.9%) saline, totaling 250 mL, over a 60minute period using a programmable pump.
  Arms: Part 1: Single Ascending Dose Escalation GC4702
Other: Placebo Dry Powder — Product matches appearance of the GC4702 dry powder formulation. The Placebo will be 500 mg Miglyol 812 oil containing up to 1% of colloidal silicon dioxide in size 1 capsule.
  Arms: Part 1: Single Ascending Dose Escalation GC4702
Other: Placebo lipid suspension — Product matches appearance of the GC4702 lipid suspension formulation. The Placebo will be 500 mg Miglyol 812 oil containing up to 1% of colloidal silicon dioxide in size 1 capsule.
  Arms: Part 1: Single Ascending Dose Escalation GC4702
Other: Fed Condition — with 240 mL (8 fluid ounces) of tap water following a high calorie/high fat meal. Subjects assigned to the fed condition will receive a standard meal per U.S. FDA guidelines7 consisting of high calorie/high fat meal prior to dosing consisting of total calories of 800-1000 of which 150, 250 and 500-600 calories are from protein, carbohydrate and fat, respectively.
  Arms: Part 2: Food Effect Study
Other: Fasting Condition — For the fasting condition, GC4702 will be administered following an overnight fast of at least 10 hours, with 240 mL (8 fluid ounces) of water. No food will be allowed for at least 4 hours post-dose. Water will be allowed as desired except for one hour before and after drug administration.
  Arms: Part 2: Food Effect Study
Drug: GC4702 lipid suspension - Part 2 — Two single doses of GC4702 (dose level to be selected based on Part 1 results), separated by a 7-day washout period
  Arms: Part 2: Food Effect Study

SUMMARY:
A Phase 1 study will test the safety, tolerability and pharmacokinetics of a single dose of GC4702 when given as an oral tablet. This study will compare capsules containing a dry powder or gel suspension of GC4702 when given orally to a similar drug called GC4419 which will be given as an intravenous infusion. This study will also assess the effect of food on the GC4702 effects.

DETAILED DESCRIPTION:
The study will be conducted in two parts: Part 1, the main study, will be a double-blind, randomized, placebo-controlled, single-ascending dose assessment of GC4702. Part 2, which will be conducted only after Part 1 and contingent upon results from Part 1, will include a food-effect cohort using a randomized design of fed/fasted conditions.

Consenting subjects will undergo screening procedures within 28 days of the start of dosing. Pharmacokinetics (PK) (parent drug and major metabolites) will be assessed in plasma and urine from all subjects.

Part 1: GC4702 or matched placebo will be administered once by mouth for a single dose. Subjects in Cohort 3 will receive a dose of (dry powder formulation) oral GC4702 48 hours after a single dose of IV GC4419 administered over 60 minutes, and a dose of (lipid suspension formulation) GC4702 one week later. Subjects in Cohorts 4 will receive a single dose of (lipid suspension formulation) oral GC4702 48 hours after a single dose of IV GC4419 administered over 60 minutes. The first 8 Subjects in Cohort 4 are dosed as required by GTO-001 Protocol Amendment 1. Upon approval of GTO-001 Protocol Amendment 2, the first 8 previously dosed Subjects (fasted with water only) are considered dosing arm 4a for the analysis, and this and subsequent cohorts become eligible for expansion to study to other dosing conditions. Cohort 4 and up will receive a single dose of IV GC4419 on Day 1 administered over 60 minutes, followed by a single dose of (lipid suspension formulation) oral GC4702 48 hours after IV dosing, under varying and distinct GC4702 dosing conditions per dose level. At discretion of Medical Monitor and upon agreement by the Principal Investigator based on available data, up to 4 arms may be evaluated, where GC4702 doses are fixed within the cohort, but oral intake conditions are modified as described below:

1. with 240 mL (8 fluid ounces) of tap water only
2. with 240 mL (8 fluid ounces) of tap water following a high calorie/high fat meal. Subjects assigned to the fed condition will receive a standard meal per U.S. FDA guidelines consisting of high calorie/high fat meal prior to dosing consisting of total calories of 800-1000 of which 150, 250 and 500-600 calories are from protein, carbohydrate and fat, respectively. For the fed condition, GC4702 will be administered following an overnight fast of at least 10 hours. Subjects will start the standard meal 30 minutes prior to administration of GC4702, and will be instructed to eat the meal in 30 minutes or less; however, the GC4702 will be administered 30 minutes after the start of the meal, with 240 mL (8 fluid ounces) of water. No food will be allowed for at least 4 hours post-dose. Water will be allowed as desired except for one hour before and after GC4702 administration. Subjects will receive standardized meals scheduled at the same time in each period of the study.
3. with 240 mL (8 fluid ounces) of orange juice only
4. with 240 mL (8 fluid ounces) of tap water, immediately followed by a single unit adult dose of the over-the-counter antacid Rennie® only Subjects will be assigned to available arms (i.e., not all arms may be tested at every cohort), and dosing arms may be evaluated concurrently, or in sequence, both considerations determined by the Medical Monitor and Principal Investigator as warranted by available data and resources.

Two forms of the oral GC4702 drug product will be tested; both formulations will be enteric-coated Capsugel Vcap Plus hard gel capsule containing (1) a dry powder formulation or (2) lipid suspension formulation.

It is anticipated that a total of 6-7 dose cohorts will be tested, including the first two dose cohorts receiving only a single oral dose of escalating doses of the encapsulated dry powder GC4702 formulation, the third cohort receiving a single oral dose of each of oral GC4702 formulation sequentially after a single IV dose of GC4419, and 3-4 subsequent cohorts receiving a single oral dose of escalating doses of the oral encapsulated lipid suspension GC4702 formulation after a single IV dose of GC4419. Depending on safety and PK results, additional cohorts may be added with either drug product preparation. See below for an overview of study design.

The first two cohorts of subjects will receive only the encapsulated dry powder formulation, to assess acute safety and oral absorption of GC4702. Six subjects will be enrolled in each of the first two cohorts, randomized 4:2 to active GC4702 or matched placebo. After each of these two cohorts, safety data will be reviewed by the internal Galera Therapeutics, Inc. (Galera) study team before proceeding to the next cohort.

The third cohort of subjects will receive both oral formulations of GC4702, sequentially, after an initial single dose of IV GC4419, to permit intra-subject assessment of the bioavailability of both formulations of GC4702. Pending initial safety and PK results in this cohort, subsequent single dose escalation is anticipated in serial cohorts receiving only the encapsulated lipid suspension formulation of GC4702 by a single dose, after an initial single dose of IV GC4419.

For cohort 3 and 4 (Amendment 1), 8 subjects per cohort will be enrolled, randomized 6:2 to active GC4702 or matched placebo.

For expansion Cohort 4 (Amendment 2), 5 and up, 8 subjects per dosing arm will be enrolled, randomized 6:2 to active or matched placebo. Assignment of Subjects to open dosing arms is at the discretion of the investigational site, which considers Subject availability, the number of dosing arms tests (1 - 4 arms per cohort), and the sequence in which each arm is evaluated with the cohort. Subject crossover to other arms is prohibited at any time, once GC4702 has been administered.

All subjects enrolled in these cohorts will first receive IV GC4419. After each of these cohorts, safety and PK data will be reviewed by the internal Galera study team before proceeding to the next cohort. Depending on the inter-subject variability in oral bioavailability, additional subjects may be added to one or more dosing cohorts.

Sentinel cohorts will be enrolled for Cohorts 1 and 3 and will be observed for 24 hours after each dose of GC4702, with safety data reviewed by the treating investigator, before additional subjects receive the scheduled dose of GC4702 in the relevant cohort. Subjects in the single-ascending dose portion of the study will also undergo electrocardiogram (ECG) monitoring at selected PK time points, to include the estimated Tmax, (anticipated to be 2-4 hours after a dose of GC4702), to assess the relationship between drug exposure to GC4419/GC4702 and effects on the QT interval.

Part 2: After completion of the single-ascending dose portion of the study, a separate cohort of subjects will receive a single dose of GC4702 (at a dose no higher than previously found to have an acceptable safety profile), with one of the oral drug products, under fasted or fed conditions, followed, after a 7-day washout period, of a second single dose of oral GC4702, at the same dose as before, under the opposite condition (fed or fasting). In the food effect cohort, subjects will be randomly assigned 1:1 to the fed-fasted sequence (i.e., either fed-first or fasted-first). For the fed condition, subjects will receive a standard meal. There will be no placebo dosing or IV GC4419 dosing in the food effect cohort

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women, age 18 and 50 years
2. Body Mass Index (BMI) 18 to 32 kg/m2, and weighing at least 50 kg at screening.
3. Blood pressure and heart rate within normal limits
4. Non-lactating, non-pregnant female, confirmed by urine pregnancy screening and willing to use acceptable methods of birth control, per medical and institutional practice.

Exclusion Criteria:

1. History of any chronic disease; or significant medical condition within three months, including but not limited to human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
2. Use of any prescription or over-the-counter medication within one week prior to baseline
3. Anticipated need for any medication during the course of the study, with the exception of contraceptive and hormone replacement therapy
4. Use of any medications that at risk for causing a precipitous decrease in blood pressure, (e.g., nitrates or erectile dysfunction drugs, from 24 hours prior to screening and throughout participation in the study)
5. Use of any vitamin or mineral supplement 24 hours prior to dosing, or anticipated use of any vitamin or mineral supplement throughout the duration of the study;
6. History of substance abuse, drug addiction, or alcoholism within 3 years prior to Baseline and/or the inability to abstain from alcohol, or drug use from 48 hours prior to the administration of study drug and throughout the duration of the study as confirmed by toxicology screens during Screening and at Baseline
7. History of smoking or any use of a tobacco product within six months prior to Baseline and/or the inability to abstain from tobacco or caffeine use from 48 hours prior to the administration of study drug and throughout the duration of the study.
8. Donation of blood or blood products within 30 days prior to the Baseline
9. Subject has previously participated in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Laboratory Abnormalities | From randomization through 4 days post last dosing in Active Phase of each cohort.
  Number of Participants With Treatment-Emergent Adverse Events and/or Laboratory Abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Galera Therapeutics, Inc.; Jason Lickliter, MBBS, PhD, FRACP, Principal Investigator — Nucleus Network; David Fuller, MD, Study Director — Syneos Health
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168